CLINICAL TRIAL: NCT01382433
Title: Clinical Assessment of Negative Symptoms Neurocognitive and Electrophysiological Characteristics in Chronic Cannabis Users
Brief Title: Chronic Cannabis Users: A Model for Negative Symptoms in Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0010-11-SHA
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Cannabis Users; Healthy Subjects
Keywords: Chronic Cannabis Users; negative symptoms; cognitive electrophysiology functions
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chronic Cannabis Users (Experimental)
  Interventions: Procedure: Magnetoencephalograph (MEG); Behavioral: Cambridge Neuropsychological Test Automated Battery (CANTAB).; Behavioral: Experimental: Scale for the Assessment of Negative Symptoms (SANS) and the Positive and Negative Syndrome Scale (PANSS)
- Control (Experimental): Neurotypical subjects
  Interventions: Procedure: Magnetoencephalograph (MEG); Behavioral: Cambridge Neuropsychological Test Automated Battery (CANTAB).; Behavioral: Experimental: Scale for the Assessment of Negative Symptoms (SANS) and the Positive and Negative Syndrome Scale (PANSS)

INTERVENTIONS:
Procedure: Magnetoencephalograph (MEG) — Brain imaging device that records the magnetic fields in the brain.
Behavioral: Cambridge Neuropsychological Test Automated Battery (CANTAB). — the CANTAB is sensitive to cognitive changes caused by a wide range of Central Nervous System disorders and medication side-effects . The CANTAB uses a computer with a touch screen, and affords a rapid and non-invasive assessment of cognitive functions.
Behavioral: Experimental: Scale for the Assessment of Negative Symptoms (SANS) and the Positive and Negative Syndrome Scale (PANSS) — The SANS and PANSS scales asses the presence and severity of Positive and Negative of Schizophrenia

SUMMARY:
The aim of the current study is set out to find a human model for negative symptoms based on clinical observation that chronic cannabis users express negative symptoms and characterize by the same neurocognitive and electrophysiology characteristics like patient suffer from schizophrenia. Towards that end the first part of the study is set out to explore weather chronic cannabis user's express negative symptoms similar to patient suffer from schizophrenia. The second part of the study will explore the neurocognitive and electrophysiology characteristics of those cannabis users that express negative symptoms. This data will be compared to parallel data of schizophrenia patients with predominantly negative symptom.

Several lines of biological and genetic evidence support the cannabinoid hypothesis for schizophrenia. Particularly, it is most significant clinically that the possible involvement of the cannabinoid system in the neural basis for the negative symptoms. This hypothesis based on clinical findings that chronic cannabis use causes a combination of symptoms including apathy, avolition, lack of interest, passivity, and cognitive impairments, the so-called "amotivational syndrome," which resembles the core negative symptoms of schizophrenia in behavioral level as well as the brain level. Both are associated with the functions or integrity of the frontal lobe due to its role in creating self-directed behaviors, deficits in which may underlie alogia, anhedonia, and flat affect. Despite the aforementioned similarities, to date, there is no documentation for such a relationship. Recognition that chronic cannabis users share the same or similar constellation of symptoms and similar neurocognitive and electrophysiology characteristics could provide a key to develop a human model for negative symptoms and an essential tool to comprehensive understanding of the etiology of negative symptoms and development of an innovative therapy.

The investigators Hypothesize That Chronic Cannabis Users Would Express the Same Constellation of Behaviors as Negative Symptoms of Schizophrenia; as well as similar neurocognitive and electrophysiology characteristics

ELIGIBILITY:
Inclusion Criteria for both groups:

1. Healthy men and women
2. Ages 20-65
3. Give informed consent for participation in the study.

Inclusion Criteria for the control:

-Used cannabis maximum 50 times in their lives, and no more than once during the past year.

Inclusion Criteria for the experimental:

-Use of cannabis for at least 2 years and in the last 6 months for at least 4 days a week.

(-After minimum 12 hours of abstinence (in order to eliminate acute cannabis effects, minimize the withdrawal effect while retaining neurophysiological effects from altered CB1 activity).

Exclusion Criteria for both groups:

(To prevent MEG artifacts by non relevant electric interference or brain conditions)

* History of epilepsy, seizure, or hot spasm, sever head injuries.
* History of metal in the head (outside the mouth space).
* History of surgery including metal implant or history of metal particles in the eye, pacemaker, or any other medical pump.
* History of migraines.
* History of drug or alcohol abuse during the last year. Inability to achieve satisfying level of communication with the subject Control Group (healthy Subjects)
* History of psychiatric diagnosis
* Drug or alcohol addiction in the year prior to the study
* History of epilepsy, seizure, or hot spasm.
* History of head injuries.
* History of metal in the head (outside the mouth space).
* History of surgery including metal implant or history of metal particles in the eye, pacemaker, or any other medical pump.
* History of migraines.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Clinical Measure | 30 min
  All participants will be assessed for negative symptoms using the Scale for the Assessment of Negative Symptoms (SANS) and the Positive and Negative Syndrome Scale (PANSS)
Cognitive Measure | 1 hour
  Cognitive Measure - All participants will be assessed for Cognitive function using the Cambridge Neuropsychological Test Automated Battery (CANTAB).
Electrophysiological Measure | 1 hour
  Electrophysiological Measure- - All participants will be assessed for Electrophysiological assesment using the MEG (Magnetoencephalogram)

CONTACTS AND LOCATIONS:
Overall Officials: Hilik Levkovitz, prof., Principal Investigator — shalvata MHC
Locations (1):
- Bar-Ilan University, Givat Shmuel, Israel